CLINICAL TRIAL: NCT00951795
Title: Clinical Evaluation of the Accuracy of the Pima™ CD4 Test for Enumeration of CD4+ T-Cell Counts
Brief Title: Accuracy of the Pima™ CD4 Test for Enumeration of CD4+ T-Cell Counts
Status: Withdrawn | Type: Observational
Sponsor: Abbott RDx Cardiometabolic (Other)
Collaborators: Inverness Medical Innovations (Industry)
Responsible Party: Meghan Bigelow (Clinical Trial Manager), Inverness Medical Innovations
Other Study IDs: BSTE-0510
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: HIV Infection; AIDS; HIV Infections
Keywords: HIV; AIDS; CD4
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adults: Adult men and women over age of 18
- Pediatrics: Pediatric boys and girls ages 12-18

SUMMARY:
This is a multi-center study designed to assess the accuracy of Pima™ CD4 Test to enumerate CD4+ T-cells in whole blood over the measurement range expected for the intended population. The Pima CD4 Test consists of the Pima™ CD4 cartridge and Pima™ Analyzer to identify and determine the absolute counts of mature helper (CD3+/CD4+) T-lymphocytes in whole blood.

DETAILED DESCRIPTION:
Blood samples will be collected from HIV infected adolescents and adult men and women presenting to a physician's office or outpatient clinic. Capillary whole blood samples will be obtained by fingerstick in duplicate from all Subjects in the study for immediate measurement of CD4+ T-cell count on the Pima CD4 Test by a trained healthcare professional. Venous whole blood samples from all Subjects in the study will also be collected and transported to the clinical laboratory of each study site for concurrent testing on the reference method by a trained laboratory professional. Venous samples from all Subjects in the study will also be measured on the Pima CD4 Test at the study site. Hematocrit will also be measured for all Subjects.

ELIGIBILITY:
Inclusion Criteria:

1. 12 years of age or older
2. Confirmed HIV infection, HIV-1 or HIV-2 according to medical history (this inclusion will be waived for healthy non-HIV infected individuals who may need to be enrolled in order to fill the high end of the CD4+ T-cell measurement range of the Pima CD4 Test.
3. Subject agrees to complete all aspects of the study

Exclusion Criteria:

1. Subject has already participated in this study at a previous date
2. Subject is enrolled in a study to evaluate a new drug
3. Patient unable or unwilling to provide informed consent
4. Vulnerable populations as deemed inappropriate for study by site principal investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The intended study population is individuals with confirmed diagnosis of HIV infection ≥ 12 years of age presenting to a physician's office or outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2009-09 (Estimated); Study Completion 2009-09

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Fenway Community Health, Boston, Massachusetts
  - University of North Carolina, Chapel Hill, North Carolina
  - Miriam Hospital, Providence, Rhode Island